CLINICAL TRIAL: NCT03403764
Title: Consciousness Field Project: Intention Host Device-mediated Distant Intentionality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merraki Institute (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Dr. Gabriele Hilberg, PhD, MFT, Principal Investigator, Merraki Institute
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 001
Record Dates: First submitted 2017-11-19; First posted 2018-01-19 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Wellness
Keywords: Intention; Distant Healing; Wellness; Distant Intentionality; Distant Healing Intention

STUDY DESIGN:
Intervention Model Description: Participants receive one of two alternative interventions during the initial phase of the study and receive the other intervention during the second phase of the study and are evaluated in parallel against a control group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigator and participants involved in this clinical trial are prevented from having knowledge which intervention is assigned to individual participants. A second control group has no knowledge of the parallel conducted Consciousness Field Project.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wellness Intention Transmission Groups (Experimental): Aim of this part of the study is to examine whether intention broadcasted from an Intention Host Device (a device which stores and transmits an intention) will affect self-compassion, general wellness, and awakening. 300 trial participants will be randomly allocated to 1/3 in control and 2/3 in the experimental IHD group, respectively. Differences in outcomes between control and experimental groups are expected.
  To address potential bias, those who enter the study but drop out are compared to those who complete the study to gauge potential differences between the two groups, and will report on this potential bias in the published manuscript.
  Interventions: Other: Wellness Intention
- Independent Control Group (No Intervention): Due to the "global, emergent entanglement" phenomenon, the investigators are curious if the investigators can test this idea within the context of the proposed study. The investigators added an additional but smaller control group which will complete the same three questionnaires for the first 6 months only and will be unaware of the larger study being conducted. These 50 subjects will be told they are completing the questionnaires in the context of a distinct, separate study and will be unaware of the Consciousness Field Project.

INTERVENTIONS:
Other: Wellness Intention
  Other Names: Distant Intentionality
  Arms: Wellness Intention Transmission Groups

SUMMARY:
This study evaluates the potential for a new kind of wellness improvement intervention, utilizing the cutting edge model of William Tiller, PhD, material scientist and Stanford Professor Emeritus. The Tiller model suggests that through the use of focused human intentionality, the investigators can impact many things, one of which is the wellness of a population. Prof. Tiller's research found that intention in the form of information can be imprinted on a simple electric device, called an Intention-Host Device, or IHD. This device then energetically broadcasts (or transmits) this information to the study participants. This present study examines what effect an intention broadcasted from an IHD has on well defined outcome variables in adult subjects, namely self-compassion, wellness, and awakening in adults.

DETAILED DESCRIPTION:
Aim of this study is to examine whether intention broadcasted from an Intention Host Device (a device which stores and transmits an intention) will affect self-compassion, general wellness, and awakening. Approximately 300 trial participants will be randomly allocated to equal groups of 1/3 in control and 2/3 in the experimental IHD group, respectively. Differences in outcomes between control and experimental groups are expected. Moreover, investigators and study participants will be blinded as to the allocation of participants.

Participants in the experimental group will receive the information from the intention broadcast for 12 consecutive months, whereas the control condition will receive no treatment for the first 6 months. After the 6-month period, the subjects allocated to the control group will begin to receive treatment in the form of the intention broadcast. To evaluate if treatment gains are sustained past the 12-month intervention period, subjects in the treatment group will provide two follow up assessments at months 15 and 18.

The first six months will enable the investigators to identify any differences in effects between the control and treatment groups. The final six months with the treatment group off the broadcast will enable the study to track the persistence of, or degradation of, any effects. Both groups will have funded 12 months of broadcast, which they will respectively receive, however in a staggered fashion. Participants will not know which group they are in until after the study and will be treated the same throughout.

Random allocation of participants will minimize known and unknown confounding variables between treatment and control group and increase likelihood of one population being studied. Attrition will pose a challenge for this longitudinal design and drop out rate is conservatively estimated to be 25%. The investigators anticipate needing to recruit and enroll approximately 300 subjects in order to attain our goal of 200 - 225 participants with complete data. With 100 subjects in each group, the investigators are expecting to 95% power (2-sided alpha 0.05, effect size d=0.5). The power estimate for this study was based on a prior IHD study by Cindy Reed which was an IRB approved study conducted at Holos University (see references). In that project, of 1784 participants invited to participate in the study nationwide, 452 began the study (took the pre-test) and 303 completed (took the post test), thus an attrition rate of 32%. The investigators anticipate less attrition in this study because of the regular teleconferences that will be offered to both the treatment and control groups.

In addition, to address potential bias, the sub-investigator, Paul Mills, Ph.D., will conduct an analysis comparing the outcomes of those who enter the study but drop out as compared to those who complete the study to gauge potential differences between the two groups, and will report on this potential bias in the published manuscript.

Primary Outcomes. Two primary outcome instruments will be used to determine treatment effects:

1. Self-Compassion Scale - Short Form (12 times). Self-compassion involves being kind toward oneself in times of pain or failure; perceiving one's experiences as part of the larger experience; and holding painful thoughts and feelings in balanced awareness. Questions are rated on a Likert scale from 1 (almost never) to 5 (almost always) with the total score derived by adding the means of each subscale together. The 6 subscales measure an individual's level of self-kindness, self-judgment, common humanity, isolation, mindfulness and over-identification.
2. PROMIS® Global Health Short Form (10 items). The 10 global health items include ratings of the five core PROMIS domains. It includes the most widely used self-rated health item (global01). PROMIS® includes a single item that provides a pure rating of physical health (global03) and another item for mental health (global04). Also included is an overall quality of life item (global02). The remaining items provide global ratings of physical function (global06), fatigue (global08), pain (global07), emotional distress (global10), and social health (global05 and global09). The 10 PROMIS® Global Health items each have 5 response choices, with the exception of the common 11-point pain intensity item ("How would you rate your pain on average" with 0=No pain and 10=Worst imaginable pain).

The treatment group and control group will be analyzed within and across subjects within the Neff Self-Compassion Scale and the PROMIS® Global Health and for emotionally meaningful expressions in their monthly online free-text testimonials. Significant pre- and post differences will be identified using the Linguistic Inquiry and Word Count (2007) text analysis software, with significance analyzed using a set of statistical tests.

Exploratory Outcome. One exploratory outcome instrument will be used to determine treatment effects: Barrett Values Inventory offers additional, exploratory data related to the spiritual growth in the participants. This inventory requires participant's selection of 10 values from a set of 40 values and will be taken every three months. Based on the participant's selections, the inventory quantitatively and qualitatively maps their psychological development across 7 dimensions (surviving, conforming, differentiating, individuating, self-actualizing, integrating, and serving). Based on how the selection of values shifts, the investigators will track the participants' progression. This assessment instrument has been used globally to map the values of individuals, organizations, communities and nations. The measurement and tracking of these outcomes will be facilitated by the Barret Values Centre, overseen by the principal investigator. The Barrett model and tools have not gone through a rigorous scientific validation process, and for this reason the basis of the study will be the two prior outcomes, with this set of outcomes being more exploratory. Because the survey template is not standardized the usual validity tests do not apply. The objective of this study is not to validate the Barrett Value Inventory but rather provide an additional exploratory data for the study.

The primary outcome instruments will be completed by participants in or around January/February of 2016 and at the end of each month thereafter until the end of the study. The exploratory Barrett instrument will be completed quarterly. Participants will be alerted during the last week of each month that forms are due on the 5th of the following month.

In addition to this stated design, the research team is interested in the purported phenomenon of "quantum entanglement" as a process that occurs between people and explains anomalous phenomena such as healing (see references). Included in this theory is the "global, emergent entanglement" phenomenon and the investigators are curious if the investigators can test this idea within the context of the proposed study. Thus, the investigators will add an additional but smaller control group which will complete the same three questionnaires for the first 6 months only and will be unaware of the larger study being conducted. These 50 subjects will be told they as subjects are completing the questionnaires in the context of a distinct, separate study and will be unaware of the Consciousness Field Project.

Outcomes. Four outcome instruments will be used to determine treatment effects:

1. Self-Compassion Scale - Short Form (12 items). Self-compassion involves being kind toward oneself in times of pain or failure; perceiving one's experiences as part of the larger experience; and holding painful thoughts and feelings in balanced awareness. Questions are rated on a Likert scale from 1 (almost never) to 5 (almost always) with the total score derived by adding the means of each subscale together. The 6 subscales measure an individual's level of self-kindness, self-judgment, common humanity, isolation, mindfulness and over-identification.
2. PROMIS® Global Health Short Form (10 items). The 10 global health items include ratings of the five core PROMIS domains. It includes the most widely used self-rated health item (global01). PROMIS® includes a single item that provides a pure rating of physical health (global03) and another item for mental health (global04). Also included is an overall quality of life item (global02). The remaining items provide global ratings of physical function (global06), fatigue (global08), pain (global07), emotional distress (global10), and social health (global05 and global09). The 10 PROMIS® Global Health items each have 5 response choices, with the exception of the common 11-point pain intensity item ("How would you rate your pain on average" with 0=No pain and 10=Worst imaginable pain).
3. Linguistic Inquiry and Word Count (2007) text analysis of emotionally meaningful expressions in participant monthly testimonials.
4. Barrett Values Inventory offers additional, exploratory data related to the spiritual growth in the participants. This inventory requires participant's selection of 10 values from a set of 40 values and will be taken every three months. Based on the participant's selections, the inventory quantitatively and qualitatively maps their psychological development across 7 dimensions (surviving, conforming, differentiating, individuating, self-actualizing, integrating, and serving). Based on how the selection of values shifts, the investigators will track the participants' progression. This assessment instrument was created in 1998 by Richard Barrett & Associates and has been used globally to map the values of individuals, organizations, communities and nations. The measurement and tracking of these outcomes will be facilitated by the Barret Values Centre, overseen by the principal investigator. The Barrett model and tools have not gone through a rigorous scientific validation process, and for this reason the basis of the study will be the two prior outcomes, with this set of outcomes being more exploratory. Because the survey template is not standardized the usual validity tests do not apply. The objective of this study is not to validate the Barrett Value Inventory but rather provide an additional exploratory data for the study.

ELIGIBILITY:
Inclusion Criteria:

* volunteers over age 18 speaking English

Exclusion Criteria:

* Subjects who cannot read, anybody with a legally authorized representative (LAR), site/sponsor employees directly involved with the study and their family members, site/sponsor employees NOT directly involved with the study and their family members, statutory minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Neff Self-Compassion Scale - Short Form | 18 months
  The Neff Short Form consists of 12 questions cover Self-Kindness (2, 6), Self-Judgment (11, 12), Common Humanity (5, 10), Isolation (4, 8), Mindfulness (3, 7), Over-Identification (1, 9) and they are rated on a Likert scale from 1 (almost never) to 5 (almost always) with the total score derived by adding the means of each subscale together. The 6 subscales measure an individual's level of self-kindness, self-judgment, common humanity, isolation, mindfulness and over-identification. Sub scale scores are calculated as the mean of the sub scale items. The total self-compassion score reverses the negative sub scale items of self-judgment, isolation, over-identification (i.e. 1=5, 2=4, 3=3, 4=2, 1=5) to compute a total mean. Change from baseline for total and subscales are tracked. Higher scores indicate higher self-compassion
NIH PROMIS Global Health Short Form | 18 months
  PROMIS® Global Health Short Form (10 items). The 10 global health items include ratings of the five core PROMIS domains. It includes the most widely used self-rated health item (global01). PROMIS® includes a single item that provides a pure rating of physical health (global03) and another item for mental health (global04). Also included is an overall quality of life item (global02). The remaining items provide global ratings of physical function (global06), fatigue (global08), pain (global07), emotional distress (global10), and social health (global05 and global09). The 10 PROMIS® Global Health items each have 5 response choices, with the exception of the common 11-point pain intensity item ("How would you rate your pain on average" with 0=No pain and 10=Worst imaginable pain). Global 1-5, 9 range from 5 (Excellent) to 1 (Poor), with higher numbers meaning greater health. Certain items are restored (Global 7 such that 5=0 no pain, and 1=10 worst pain), Global8 (5=None, 1=Very Severe),

SECONDARY OUTCOMES:
The text analysis Linguistic Inquiry and Word Count (2007) | 18 months
  Linguistic Inquiry and Word Count (2007) performs quantitative text analysis of freeform participant survey comments across a variety of content categories like emotion, affect, social, personal concern, biological processes, tone. The percentage of words in content categories will be tracked over time for increase in occurrence of positive categories and a decrease in occurrence in negative categories during broadcast relative to non-broadcast periods.
Barrett Values Inventory | 18 months
  Barrett Values Inventory offers additional, exploratory data related to the psychological and spiritual growth in the participants. This inventory requires participant's selection of 10 values from a set of 40 values and will be taken every three months. Based on the participant's selections, the inventory quantitatively and qualitatively maps their psychological and spiritual development across 7 dimensions (surviving, conforming, differentiating, individuating, self-actualizing, integrating, and serving). Based on a shift in the selection of values, the investigators will track the participants' progression through these 7 levels, with progression over time from Levels 1-3 (ego-based values) to Level 4 (individuation - facing change) and rising Levels 5-7 (spiritual values) being expressed as positive.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mills, Ph.D., Study Director — Professor of Family Medicine and Public Health, UC San Diego
Locations (1):
- Merraki Institute, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Radin D, Hayssen G, Walsh J. Effects of intentionally enhanced chocolate on mood. Explore (NY). 2007 Sep-Oct;3(5):485-92. doi: 10.1016/j.explore.2007.06.004. PMID 17905358
- [Background] Radin D, Schlitz M, Baur C. Distant Healing Intention Therapies: An Overview of the Scientific Evidence. Glob Adv Health Med. 2015 Nov;4(Suppl):67-71. doi: 10.7453/gahmj.2015.012.suppl. Epub 2015 Nov 1. PMID 26665044
- [Background] Targ E. Evaluating distant healing: a research review. Altern Ther Health Med. 1997 Nov;3(6):74-8. PMID 9375432
- [Background] Nisha Manek, William Tiller. Feasibility of Information Medicine as Delivered by Intention Host Devices: A Case Report Glob Adv Health Med. 2013 Nov; 2(Suppl): S152. Published online 2013 Nov 1. doi: 10.7453/gahmj.2013.097CP.P05.09 PMCID: PMC3875095
- [Background] Hyland ME. Does a form of 'entanglement' between people explain healing? An examination of hypotheses and methodology. Complement Ther Med. 2004 Dec;12(4):198-208. doi: 10.1016/j.ctim.2004.10.002. PMID 15649833
- See also: Whitepapers: #1 and # XVI and # XXIV and # XXX and # XXI — http://Tiller.org